CLINICAL TRIAL: NCT07074899
Title: Development and Evaluation of a Multi-Component Intervention to Support HIV Testing and Linkage to Services Among Men Who Have Sex With Men (MSM) in Perú ("PROJECT MERCURY")
Brief Title: Evaluation of a Multi-Component Intervention to Support HIV Testing and Linkage to Services Among MSM in Peru
Acronym: MERCURY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Asociación Civil Via Libre, Peru (Other); Epicentro, Peru (Unknown)
Responsible Party: Principal Investigator, Alexander Lankowski, MD, Associate in VIDD, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RG1121536; K23MH126781 (NIH); FHIRB0010738 (Other: Fred Hutchinson Cancer Center IRB)
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Mobile Health; Feasibility Studies; Qualitative Research; Implementation Science; Social Determinants of Health; Health Services Accessibility; Global Health; HIV Prevention; HIV Testing; Linkage to Care
Keywords: HIV self-test; HIV prevention; Latin America; Linkage to care; Community-based HIV testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Mercury

STUDY DESIGN:
Intervention Model Description: Intervention arm is randomly assigned at the level of the recruitment date.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Rapid Test (Active Comparator): Participants will receive a rapid HIV test on-site at the time of enrollment.
  Interventions: Other: Multi-component HIV testing and linkage-to-services intervention
- Group 2 - HIV Self-Test (Active Comparator): Participants will be given an HIV self-test kit that they may use at the time and place of their choosing.
  Interventions: Other: Multi-component HIV testing and linkage-to-services intervention
- Group 3 - Coupon (Active Comparator): Participants will be given a coupon redeemable for a free future HIV test at a participating health center.
  Interventions: Other: Multi-component HIV testing and linkage-to-services intervention
- Group 4 - "Choice" (Active Comparator): Participants will be offered their choice of any one of the three HIV testing formats (rapid test, self-test, referral coupon).
  Interventions: Other: Multi-component HIV testing and linkage-to-services intervention

INTERVENTIONS:
Other: Multi-component HIV testing and linkage-to-services intervention — The intervention includes two core components:
  1. HIV testing offered at sex-on-premises-venues [SOPVs];
  2. mHealth-supported linkage to treatment/prevention services (enrollment in a two-way text messaging application adapted from the WelTel platform).
  In this trial, the specific format of HIV testing offered will differ according to intervention arm.
  Other Names: Mercury

SUMMARY:
This study is testing a new program designed to improve access to HIV testing and help connect people with available treatment or prevention services, based on their test result. The version of the program being tested in this study was designed for men who have sex with men (MSM) in Lima, Peru. The program has two main parts: 1) offering HIV testing at venues where people go for sex (called "sex-on-premises venues" or SOPVs), and 2) a text messaging app that shares useful information about HIV treatment/prevention; users can also message back to get support from a healthcare worker. Before doing this study, the researchers worked with community members and healthcare providers in the area to make sure that the HIV testing approach and mobile app were designed in a way that would be engaging and meet their needs.

Every Thursday, Friday, and Saturday night during recruitment, the researchers will go to SOPVs popular among the MSM community in Lima and invite people to take an HIV test. On each recruitment date, they will offer one of the following HIV testing options:

1. A rapid HIV test done on-site (participants will get their result right away)
2. An HIV self-testing kit to take home
3. A coupon for a free HIV test at a participating health center
4. Their choice of any one of the previous three options

Only one of these options will be offered at a time, depending on the date. The specific HIV testing option offered on each date will be randomly assigned. All participants will receive the mobile app, which will send weekly messages with links to different types of online content (infographics, maps, videos) over the next 3 months. The specific sequence of messages and content will be different depending on the type of HIV test the person received and their HIV test result, once it is known.

The study will measure two main outcomes related to the acceptability and feasibility of the program:

* The number and percentage of people who accept the program when offered
* The number and percentage of participants who continue to engage with the mobile app after 3 months

The study will also measure:

* overall satisfaction with the app (based on a questionnaire sent at 3 months)
* the number and percentage of participants who completed any form of HIV testing after 3 months
* the number and percentage of participants who started HIV treatment (out of those with a positive HIV test)
* the number and percentage of participants who started HIV pre-exposure prophylaxis, or "PrEP" (out of those with a negative HIV test)

All follow-up will be done remotely. Participants will have the app for 3 months. After 3 months, they will get a follow-up questionnaire asking about their experiences with the program. The researchers will keep tracking results related to the HIV treatment/prevention services that people receive for up to 6 months.

DETAILED DESCRIPTION:
This study will evaluate the feasibility, acceptability, and preliminary effectiveness of a multi-component HIV testing and linkage-to-services intervention ("Mercury") among MSM in Lima, Peru. The Mercury intervention includes two core components: 1) HIV testing offered at sex-on-premises venues (SOPVs, e.g., saunas, hourly hotels, bars/discos with dark rooms); and 2) a mobile health (mHealth) application consisting of bidirectional SMS text messaging and tailored multimedia content related to HIV treatment/prevention and other sexual health topics.

The Mercury application is adapted from a previously validated mHealth technology platform (WelTel). In addition to its use as a system for secure two-way messaging with healthcare providers, the application is programmed to send two types of standardized weekly text messages:

* "Checkins" containing a generic greeting, phrased in the form of a question (e.g., "Hi [username], how are you?"), with user responses automatically classified ("OK", "NOT OK", or "Unrecognized") and presented in a web-based dashboard to facilitate follow-up, as needed, by the provider team
* "Topical Messages" containing links to tailored multimedia content (infographics, videos, service locator maps) based on the user's HIV testing scenario and result (HIV+, HIV-, pending HIV result).

In this randomized trial, the researchers will compare four HIV testing strategies in the context of the Mercury intervention, corresponding to the following intervention arms:

* Arm 1: Rapid HIV Test, participants will receive a rapid HIV test performed on-site at the venue.
* Arm 2: HIV Self-Test, participants will be given an HIV self-test kit to take home.
* Arm 3: Coupon, participants will receive a digital coupon redeemable for a free HIV test at one of the referral clinics affiliated with the study.
* Arm 4: "Choice", participants can choose whichever one of the three above-mentioned forms of HIV testing they most prefer.

Every Thursday, Friday, and Saturday during recruitment, the intervention will be offered at a single SOPV in downtown Lima. There will be three recruitment venues overall, which will alternate based on day of the week: SOPV#1 [Thursdays], SOPV#2 [Fridays], SOPV#3 [Saturdays]). On each given recruitment date, only one of the four HIV testing strategies (i.e., intervention arms) will be offered - assigned at random using a block randomization scheme designed to generate an even (1:1:1:1) distribution of recruitment dates by intervention arm, balanced by day of week (Thu vs Fri vs Sat) and recruitment venue (SOPV#1 vs SOPV#2 vs SOPV#3). All participants will receive the mHealth application, including tailored content related to the HIV testing format they received. The study team will approach potential participants as they enter or leave the venue, introducing the study with a brief (< 30 second) standardized script describing the HIV testing format on offer. For those who accept the intervention and enroll in the study, eligibility screening, informed consent, and receipt of the corresponding HIV testing format will be done in a private space (either inside the venue or in a secure van parked outside). All participants will receive standard HIV pre-test counseling according to Peruvian national guidelines and complete a baseline questionnaire collecting data on socio-demographics, use of mobile technology, and experience with HIV testing/prevention. There are no in-person follow-up visits as part of this study. Participants will be enrolled in the mHealth application for a total of 3 months, at which time they will be contacted by the study team and asked to complete a follow-up questionnaire. The researchers may continue to observe participants for up to 6 months, if necessary, to ascertain outcomes.

The study will evaluate two co-primary outcomes: uptake of the intervention (number who accept the intervention divided by the number offered), and continued engagement with the mHealth application (assessed at 3 months). Additionally, the following secondary outcomes will be assessed: HIV test completion, and user satisfaction with the mHealth application. Exploratory outcomes will include: linkage to care and HIV treatment initiation (if HIV+); linkage to prevention and HIV pre-exposure prophylaxis (PrEP) initiation (if HIV-).

ELIGIBILITY:
Inclusion criteria:

1. age ≥ 18 years
2. identifies as gay, bisexual, or other man who has sex with men (MSM)
3. attendance at the designated recruitment venue (SOPV) and is willing to receive the form HIV testing (i.e., intervention arm) offered on that recruitment date
4. has a mobile phone device and service capable of two-way SMS text messaging via the WelTel platform and is willing to send/receive text messages using their primary mobile phone number
5. able to read and write

Exclusion criteria:

1. self-reports having a previous HIV diagnosis
2. cognitively or psychologically unable to participate in HIV testing (e.g. visibly intoxicated or self-reports being intoxicated)
3. unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 150 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-12-13 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Uptake | 30 minutes
  The proportion of individuals who accept the intervention and enroll in the study among those who are approached and offered the intervention at the recruitment venue.
Continued Engagement | 3 months
  The proportion of participants who remain engaged with the mHealth component of the intervention over time, as indicated by having either 1) sent at least one text message reply (either responding directly to a programmed message or spontaneously messaging the provider team) or 2) logged into the WelTel online portal (or otherwise accessed the application content) within the previous 15 days.

SECONDARY OUTCOMES:
HIV test completion | 3 months
  The proportion of participants confirmed to have completed an HIV test within 3 months of enrollment.
User satisfaction | 3 months
  This will be a composite outcome based on an online questionnaire participants will be sent gauging their overall satisfaction with the mHealth component of the intervention.

OTHER OUTCOMES:
Linkage to HIV care | 3 months, 6 months
  Among participants who test HIV positive, the proportion who establish care with an HIV treatment provider (as indicated by completion of a clinic intake visit) within 3 or 6 months of their study-provided HIV test result.
ART initiation | 3 months, 6 months
  Among participants who test HIV positive, the proportion who initiate antiretroviral treatment (ART) within 3 or 6 months of their study-provided HIV test result.
Linkage to HIV prevention | 3 months, 6 months
  Among participants who test HIV negative, the proportion who establish care (as indicated by completion of a clinic intake visit) with an HIV pre-exposure prophylaxis (PrEP) provider within 3 or 6 months of their study-provided HIV test result.
PrEP initiation | 3 months, 6 months
  Among participants who test HIV negative, the proportion who initiate HIV pre-exposure prophylaxis (PrEP) within 3 or 6 months of their study-provided HIV test result.
HIV seropositivity | 6 months
  The proportion of participants with a confirmed HIV positive result on the study-provided test.
Receipt of viral load testing | 6 months
  Among participants who test HIV positive, the proportion with documentation of at least one viral load test having been performed.
PrEP attitudes, willingness and intention to use | 3 months
  Among participants who test HIV negative, the motivational PrEP cascade will be assessed using a questionnaire sent 3 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (2):
- Peru (2):
  - Epicentro, Lima, Lima Province
  - Via Libre, Lima, Lima Province

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data (baseline and follow-up surveys; primary, secondary, and exploratory outcomes) may be shared upon reasonable request by contacting the Principal Investigator.
Supporting Information: Study Protocol, ICF